CLINICAL TRIAL: NCT04182555
Title: Identification of Jaundice in Newborns Using Smartphones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Helse Fonna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/1608
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Jaundice, Neonatal; Hyperbilirubinemia, Neonatal
Keywords: Diagnosis; Cell Phones; Infant, Newborn; Skin Pigmentation
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal; Disease; Pigmentation Disorders

STUDY DESIGN:
Intervention Model Description: 200 newborns with varying degree of jaundice will be recruited.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newborns in St.Olavs Hospital and Haugesund Hospital (Experimental): All newborns will be examined through 4 different methods of determining jaundice.
  Interventions: Device: Bilirubin estimates from Smartphone Application; Diagnostic Test: Bilirubin concentration measured in standard blood samples; Device: Bilirubin estimates from standard transcutaneous device; Other: Visual assessment of jaundice

INTERVENTIONS:
Device: Bilirubin estimates from Smartphone Application — Bilirubin estimates through color analysis of digital images obtained through smartphone application.
Diagnostic Test: Bilirubin concentration measured in standard blood samples — Bilirubin measured in total serum bilirubin.
Device: Bilirubin estimates from standard transcutaneous device — Bilirubin estimates performed by transcutaneous device ( Dräger JM-105)
Other: Visual assessment of jaundice — Degree of jaundice will be assessed by Kramer scale

SUMMARY:
Neonatal jaundice is a common and most often harmless condition. However, when unrecognized it can be fatal or cause serious brain injury. Three quarters of these deaths are estimated to occur in the poorest regions of the world. The treatment of jaundice, phototherapy, is in most cases easy, low-cost and harmless. The crucial point in reducing the burden of disease is therefore to identify then children at risk. This results in the need for low-cost, reliable and easy-to-use diagnostic tools that can identify newborns with jaundice.

Based on previous research on the bio-optics of jaundiced newborn skin, a prototype of a smartphone application was developed and tested in a pilot study and the application refined.

This smartphone application will now be evaluated in a clinical trial set in two hospitals in Norway. The smartphone application gives immediate estimates of bilirubin values in newborns, and these estimates will be compared to the bilirubin levels measured in standard blood samples, as well as the results from ordinary transcutaneous measurement devices.

DETAILED DESCRIPTION:
The smartphone jaundice app system works by taking pictures of newborns with a custom-made color calibration card placed on their chest. This makes it possible to measure the skin color precisely regardless of the specific light source that is used to illuminate the newborn. The measured skin color is then compared with items in a database of simulated newborn skin colors. These simulated newborn skin colors have been created using numerical simulations of how light moves through skin, with varying skin parameters including, but not limited to, skin thickness, blood concentration, melanin, and of course bilirubin, the pigment that causes jaundice. By comparing the measured skin color with the simulated skin colors that are most similar to it, the investigators can then estimate the bilirubin concentration in the newborn's skin by e.g. averaging the bilirubin concentrations used to create these simulated skin colors.

In a group of 200 newborns with varying degree of jaundice, correlation between smartphone bilirubin estimates will be compared with total serum bilirubin and standard transcutaneous bilirubinometry.

ELIGIBILITY:
Inclusion Criteria:

* Born in St.Olavs hospital, Trondheim or in Haugesund Hospital, Norway
* Born with gestational age >36+6
* Birth weight ≥ 2500g and <4500g
* Age 1 - <15 days
* Are having a blood sample performed, as newborn screening or for jaundice assessment

Exclusion criteria:

Infants needing intensive treatment. This includes:

* Infants in the need for respiratory support
* Infants with conditions that could compromise skin circulation, as sepsis, heart failure or other
* Infants that have received phototherapy

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Smartphone application sensitivity | 5 minutes
  Sensitivity of the smartphone application to detect severe jaundice, defined as total serum bilirubin value > 250 umol/l.

SECONDARY OUTCOMES:
Repeatability | 5 min
  To evaluate the repeatability of multiple measurements with the new smartphone tool
Correlation between bilirubin estimates by smartphone pictures and by total serum bilirubin | 5 minutes
  Estimate of bilirubin levels from smartphone pictures, compared with bilirubin measurements in total serum. Correlation will be expressed by Pearson correlation coefficient, r.
Correlation between bilirubin estimates by smartphone pictures and by standard transcutaneous readings. | 5 minutes
  To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from a standard transcutaneous device in newborns with varying degree of jaundice. Correlation will be expressed by Pearson correlation coefficient, r.
Correlation between bilirubin estimates by smartphone pictures and visual assessment of jaundice | 5 min
  - To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from visual inspection in newborns with varying degree of jaundice

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, md prof, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Haugesund Hospital, Haugesund
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No